CLINICAL TRIAL: NCT03734237
Title: A Pragmatic Assessment of Influenza Vaccine Effectiveness in the DoD
Acronym: PAIVED
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency); Defense Health Agency Immunization Healthcare Branch (Unknown); US Department of Defense Armed Forces Health Surveillance Center (U.S. Federal Agency); Naval Health Research Center (U.S. Federal Agency); United States Air Force School of Aerospace Medicine (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDCRP-120; AAI1201200007000 (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2018-11-02; First posted 2018-11-07 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Influenza; Influenza-like Illness; Influenza Vaccines
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: A total of 18,000 eligible subjects (or 6,000 subject distributed evenly between the 3 study arms) will be enrolled. eligible subjects will be randomized in 1:1:1 (cell-culture-based vaccine, the recombinant vaccine, or the egg-based vaccine) over four influenza seasons (2018-2019,2019-2020, 2020-2021, and 2021-2022).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Egg based influenza vaccines (Active Comparator): Quadrivalent egg-based vaccines, which contain an inactivated form of the virus. Vaccines will be given to the participant in accordance with standard clinical practices for those in the US military. All egg-based vaccines are FDA licensed for use in the United States.
  Interventions: Biological: Egg based influenza vaccines
- Recombinant influenza vaccines (Active Comparator): FluBlok, recombinant HA influenza vaccine. Vaccines will be given to the participant in accordance with standard clinical practices for those in the US military. Flublok Quadrivalent is a quadrivalent recombinant influenza vaccine that has been licensed by the FDA for use in the United States.
  Interventions: Biological: Recombinant influenza vaccines
- Cell-culture based influenza vaccines (Active Comparator): Flucelvax, Madin-Darby canine kidney (MDCK)-cell-culture based inactivated influenza vaccine. Vaccines will be given to the participant in accordance with standard clinical practices for those in the US military. Flucelvax quadrivalent, the only cell-based flu vaccine FDA licensed for use in the United States.
  Interventions: Biological: Cell-culture based influenza vaccines

INTERVENTIONS:
Biological: Egg based influenza vaccines — Participants will be randomly allocated to one of three vaccine types in accordance with standard clinical practices for those in the US military. All vaccines are FDA licensed for use in the United States.
  Arms: Egg based influenza vaccines
Biological: Recombinant influenza vaccines — Participants will be randomly allocated to one of three vaccine types in accordance with standard clinical practices for those in the US military. All vaccines are FDA licensed for use in the United States.
  Arms: Recombinant influenza vaccines
Biological: Cell-culture based influenza vaccines — Participants will be randomly allocated to one of three vaccine types in accordance with standard clinical practices for those in the US military. All vaccines are FDA licensed for use in the United States.
  Arms: Cell-culture based influenza vaccines

SUMMARY:
A total of 18,000 eligible subjects (or 6,000 subject distributed evenly between the 3 study arms) will be enrolled. Eligible subjects will be randomized in 1:1:1 (cell-culture-based vaccine, the recombinant vaccine, or the egg-based vaccine) over four influenza seasons (2018-2019, 2019-2020, 2020-2021, and 2021-2022).

DETAILED DESCRIPTION:
This four-year, pragmatic, prospective study will compare the effectiveness of licensed egg-based inactivated influenza vaccines to the effectiveness of two other types of licensed vaccines, the cell-culture based inactivated influenza vaccine and the recombinant influenza vaccine, in the prevention of laboratory-confirmed influenza infection in active duty members, military retirees, and other DoD beneficiaries. Military treatment facilities (MTFs) in the United States will participate in this protocol. Enrollment will be restricted to adults (≥18 years and older) who are preparing to receive seasonal influenza vaccination at participating DoD sites. Subjects will be randomized to receive one of the three licensed influenza vaccines types for evaluation of effectiveness. There is no exclusion for pregnancy, as none of these licensed products are contraindicated in pregnant women.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible for care in Department of Defense medical facilities (Defense Enrollment Eligibility Reporting System eligible)
2. ≥18 years of age.
3. At a participating Military Treatment Facility site for the purpose of receiving a seasonal (2018-2019, 2019-2020,2020-2021, 2021-2022) influenza vaccination.
4. Able to speak English and able to provide informed consent
5. Able to receive and respond to texts and/or emails, or a military recruit

Exclusion Criteria:

1. Adults intending to receive or who have received the current seasons FluMist Vaccine (LAIV)
2. Adults who have already received a flu vaccine within the current season
3. Individual who cannot receive a flu vaccine or standard dosing due to another medical condition
4. Allergic to gentamicin, polymyxin and/or neomycin
5. Individuals who fail to meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15449 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2024-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Burgess, MD, Principal Investigator — Uniformed Services University of the Health Sciences; Rhonda Colombo, MD, Study Director — Infectious Diseases Clinical Research Program
Locations (9):
- United States (9):
  - Naval Medical Center San Diego, San Diego, California
  - United States Naval Academy, Annapolis, Maryland
  - USU, Bethesda, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Lackland Airforce Base, San Antonio, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - Madigan Army Medical Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez JL, Cooper MJ, Myers CA, Cummings JF, Vest KG, Russell KL, Sanchez JL, Hiser MJ, Gaydos CA. Respiratory Infections in the U.S. Military: Recent Experience and Control. Clin Microbiol Rev. 2015 Jul;28(3):743-800. doi: 10.1128/CMR.00039-14. PMID 26085551
- [Background] Flannery B, Chung JR, Belongia EA, McLean HQ, Gaglani M, Murthy K, Zimmerman RK, Nowalk MP, Jackson ML, Jackson LA, Monto AS, Martin ET, Foust A, Sessions W, Berman L, Barnes JR, Spencer S, Fry AM. Interim Estimates of 2017-18 Seasonal Influenza Vaccine Effectiveness - United States, February 2018. MMWR Morb Mortal Wkly Rep. 2018 Feb 16;67(6):180-185. doi: 10.15585/mmwr.mm6706a2. PMID 29447141
- [Background] Zost SJ, Parkhouse K, Gumina ME, Kim K, Diaz Perez S, Wilson PC, Treanor JJ, Sant AJ, Cobey S, Hensley SE. Contemporary H3N2 influenza viruses have a glycosylation site that alters binding of antibodies elicited by egg-adapted vaccine strains. Proc Natl Acad Sci U S A. 2017 Nov 21;114(47):12578-12583. doi: 10.1073/pnas.1712377114. Epub 2017 Nov 6. PMID 29109276
- [Background] Wu NC, Zost SJ, Thompson AJ, Oyen D, Nycholat CM, McBride R, Paulson JC, Hensley SE, Wilson IA. A structural explanation for the low effectiveness of the seasonal influenza H3N2 vaccine. PLoS Pathog. 2017 Oct 23;13(10):e1006682. doi: 10.1371/journal.ppat.1006682. eCollection 2017 Oct. PMID 29059230
- [Background] Skowronski DM, Janjua NZ, De Serres G, Sabaiduc S, Eshaghi A, Dickinson JA, Fonseca K, Winter AL, Gubbay JB, Krajden M, Petric M, Charest H, Bastien N, Kwindt TL, Mahmud SM, Van Caeseele P, Li Y. Low 2012-13 influenza vaccine effectiveness associated with mutation in the egg-adapted H3N2 vaccine strain not antigenic drift in circulating viruses. PLoS One. 2014 Mar 25;9(3):e92153. doi: 10.1371/journal.pone.0092153. eCollection 2014. PMID 24667168
- [Background] Cobey S, Gouma S, Parkhouse K, Chambers BS, Ertl HC, Schmader KE, Halpin RA, Lin X, Stockwell TB, Das SR, Landon E, Tesic V, Youngster I, Pinsky BA, Wentworth DE, Hensley SE, Grad YH. Poor Immunogenicity, Not Vaccine Strain Egg Adaptation, May Explain the Low H3N2 Influenza Vaccine Effectiveness in 2012-2013. Clin Infect Dis. 2018 Jul 18;67(3):327-333. doi: 10.1093/cid/ciy097. PMID 29471464
- [Background] Wang W, Butler EN, Veguilla V, Vassell R, Thomas JT, Moos M Jr, Ye Z, Hancock K, Weiss CD. Establishment of retroviral pseudotypes with influenza hemagglutinins from H1, H3, and H5 subtypes for sensitive and specific detection of neutralizing antibodies. J Virol Methods. 2008 Nov;153(2):111-9. doi: 10.1016/j.jviromet.2008.07.015. Epub 2008 Sep 4. PMID 18722473
- [Background] Wang W, Xie H, Ye Z, Vassell R, Weiss CD. Characterization of lentiviral pseudotypes with influenza H5N1 hemagglutinin and their performance in neutralization assays. J Virol Methods. 2010 May;165(2):305-10. doi: 10.1016/j.jviromet.2010.02.009. Epub 2010 Feb 11. PMID 20153374
- [Derived] Colombo RE, Richard SA, Schmidt K, Schofield C, Ganesan A, Campbell W, Hrncir D, Lalani T, Mende K, Markelz AE, Berjohn CM, Housel L, Becher D, Zell ER, Ewing D, Sundaram AK, Modi JR, Saperstein A, Tilley DH Jr, Williams A, McClenathan B, Collins L, Spooner C, Seshadri S, Fries A, Maves RC, Powers Iii JH, O'Connell RJ, Pollett SD, Simons MP, Coles CL, Burgess TH; PAIVED Study Group. Randomized Pragmatic Trial of the Comparative Effectiveness of Chicken Egg-Based Inactivated, Mammalian Cell Culture-Based Inactivated, and Recombinant Protein Quadrivalent Seasonal Influenza Vaccines in United States Military Health System Beneficiaries. Clin Infect Dis. 2025 Dec 24;81(5):e454-e463. doi: 10.1093/cid/ciaf503. PMID 40973113
- See also: Influenza. Centers for Disease Control and Prevention — https://www.cdc.gov/flu/index.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from adult military health system (MHS) beneficiaries preparing to receive a seasonal influenza vaccination at a participating DoD site. Eligible participants who provided informed consent were block randomized 1:1:1 to receive one of three types of licensed influenza vaccines (cell-culture-based vaccine, recombinant vaccine, or egg-derived vaccine). The first participant was enrolled in November 2018, and the last participant was enrolled in January 2022.
Pre-assignment Details: Among 15449 enrolled participants, 17 were excluded from analysis due to ineligibility (i.e., not eligible for care in MHS, already received an influenza vaccination, etc).
Groups:
- Egg-based Vaccine: Subjects vaccinated with egg-based vaccine.
- Recombinant Vaccine: Subjects vaccinated with recombinant vaccine.
- Cell-derived Vaccine: Subjects vaccinated with cell-derived vaccine.
Period: Overall Study
Arm/Group | Egg-based Vaccine | Recombinant Vaccine | Cell-derived Vaccine
Started | 5145 | 5150 | 5137
Completed | 5137 | 5138 | 5127
Not Completed | 8 | 12 | 10
Not completed — Lost to Follow-up | 1 | 3 | 0
Not completed — Withdrawal by Subject | 7 | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Egg-based Vaccine | Recombinant Vaccine | Cell-derived Vaccine | Total
Number analyzed (Participants) | 5145 | 5150 | 5137 | 15432
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 4944 | 4954 | 4947 | 14845
  >=65 years | 201 | 196 | 190 | 587
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1635 | 1672 | 1649 | 4956
  Male | 3510 | 3478 | 3488 | 10476
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 995 | 984 | 955 | 2934
  Not Hispanic or Latino | 4025 | 4048 | 4051 | 12124
  Unknown or Not Reported | 125 | 118 | 131 | 374
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 51 | 49 | 44 | 144
  Asian | 289 | 315 | 316 | 920
  Native Hawaiian or Other Pacific Islander | 48 | 63 | 50 | 161
  Black or African American | 600 | 643 | 606 | 1849
  White | 3575 | 3504 | 3546 | 10625
  More than one race | 281 | 270 | 284 | 835
  Unknown or Not Reported | 301 | 306 | 291 | 898
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5145 | 5150 | 5137 | 15432

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Laboratory Confirmed Influenza
Description: Laboratory-confirmed influenza as ascertained by a sensitive and specific assay.
Time Frame: Onset > 13 days after vaccination up to 1 year
Population: Analysis based on actual vaccine received.
Measure: Number; unit: participants
Arm/Group | Egg-based Vaccine | Cell-derived Vaccine | Recombinant Vaccine
Number analyzed (Participants) | 5145 | 5137 | 5150
participants | 68 | 86 | 77
Statistical Analysis 1: Comparison: Egg-based Vaccine vs Cell-derived Vaccine; Relative vaccine effectiveness with the outcome laboratory confirmed influenza identified via surveillance and/or abstracted from clinical records; Test type: Equivalence — Null Hypothesis: RR=1, Alternative hypothesis: RR not equal to 1; p = 0.1412, Chi-squared; Risk Ratio (RR) = -26.7, 95% CI 2-sided [-73.7 to 7.6]
Statistical Analysis 2: Comparison: Egg-based Vaccine vs Recombinant Vaccine; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — Null Hypothesis: RR=1, Alternative hypothesis: RR not equal to 1; p = 0.4552, Chi-squared; Risk Ratio (RR) = -13.1, 95% CI 2-sided [-56.4 to 18.2]

2. Secondary Outcome: Hemagglutination Inhibition (HI) Titer Responses to Influenza Vaccine Strains.
Description: Strain-specific seroconversion rate determined by reference hemagglutination inhibition assay.
Time Frame: Baseline to 21-35 days post vaccine
Population: Substudy participants were included if they had pre- and post-vaccination samples.
Measure: Number; unit: participants
Groups:
- Egg-based Vaccine: Subset of immunogenicity subjects vaccinated with egg-based vaccine.
- Cell-derived Vaccine: Subset of immunogenicity subjects vaccinated with cell-derived vaccine.
- Recombinant Vaccine: Subset of immunogenicity subjects vaccinated with recombinant vaccine.
Arm/Group | Egg-based Vaccine | Cell-derived Vaccine | Recombinant Vaccine
Number analyzed (Participants) | 355 | 359 | 373
participants
  H1N1: Number with 4-fold rise in HI | 103 | 114 | 184
  H3N2: Number with 4-fold rise in HI | 108 | 158 | 267
  B-Victoria: Number with 4-fold rise in HI | 49 | 48 | 92
  B-Yamagata: Number with 4-fold rise in HI | 19 | 24 | 64

3. Secondary Outcome: Pseudovirion Neutralization (PVN) Responses to Influenza Vaccine.
Description: Neutralizing antibody responses (4-fold rise) to HA-psuedoviruses corresponding to vaccine-matched viruses, recently circulating influenza virus, and emerging influenza strain.
Time Frame: Baseline to 21-35 days post vaccine
Measure: Number; unit: percentage of participants
Groups:
- Egg Based Influenza Vaccines: Subset of immunogenicity subjects vaccinated with egg-vaccine (2018-19)
- Cell-derived Vaccine: Subset of immunogenicity subjects vaccinated with cell-derived vaccine (2018-19)
- Recombinant Vaccine: Subset of immunogenicity subjects vaccinated with recombinant vaccine (2018-19)
Arm/Group | Egg Based Influenza Vaccines | Cell-derived Vaccine | Recombinant Vaccine
Number analyzed (Participants) | 46 | 36 | 51
percentage of participants
  Seroconversion rate against egg-passaged HA-pseudovirus (SGP/19/16 NIB-104) | 8.7 | 13.9 | 47.1
  Seroconversion rate against cell-passaged HA-pseudovirus (NC/04/16) | 8.7 | 8.3 | 43.1
  Seroconversion rate against wild-type (SGP/19/16; recombinant HA-pseudovirus) | 4.3 | 16.7 | 56.9
  Seroconversion rate against HA-pseudovirus corresponding to prior season vaccine strain | 6.5 | 13.9 | 62.7
  Seroconversion rate against HA-pseudovirus corresponding to recently circulating virus | 4.3 | 11.1 | 52.9
  Seroconversion rate against HA-pseudovirus corresponding to emerging infuenza strain | 2.2 | 0 | 21.6

4. Secondary Outcome: Anti-Neuraminidase (Anti-NA) Titer Responses to Influenza Vaccine.
Description: Anti-Neuraminidase (Anti-NA) titer responses determined by enzyme linked immuno-assay.
Time Frame: Baseline to 21-35 days post vaccine
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean titer
Arm/Group | Egg Based Influenza Vaccines | Cell-derived Vaccine | Recombinant Vaccine
Number analyzed (Participants) | 46 | 32 | 51
geometric mean titer
  N1 Titer, Pre-vaccination | 53.7 [41.1 to 70.1] | 121.2 [78.9 to 186.1] | 80.7 [58.4 to 111.5]
  N1 Titer, Post-vaccination | 207.1 [146.6 to 292.6] | 118.3 [76.9 to 182.1] | 77.7 [56.8 to 106.2]
  N2 Titer, Pre-vaccination | 121.2 [94.3 to 156.0] | 126.0 [82.7 to 191.8] | 83.0 [67.6 to 102]
  N2 Titer, Post-vaccination | 291.5 [216.0 to 393.2] | 230.5 [150.6 to 352.9] | 78.4 [63.4 to 96.9]

5. Secondary Outcome: Number of Participants With Influenza-Like Illness
Description: Rate of protocol defined influenza-like illness ascertained by participant response to active surveillance.
Time Frame: Onset > 13 days after vaccination up to 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Egg-based Influenza Vaccine: Subjects vaccinated with egg-based vaccine.
Arm/Group | Egg-based Influenza Vaccine | Recombinant Vaccine | Cell-derived Vaccine
Number analyzed (Participants) | 5145 | 5150 | 5137
Participants | 1055 | 1120 | 1080

6. Other Pre Specified Outcome: Number of Participants With SARS-CoV-2 and Influenza Co-Infection
Description: Laboratory-confirmed SARS CoV2, and SARS CoV2 plus influenza co-infection, as ascertained by nasal swab PCR.
Time Frame: Onset > 13 days after influenza vaccination up until one year
Population: Participants enrolled in PAIVED beginning in 2019-20 season.
Measure: Count of Participants; unit: Participants
Groups:
- Cell-derived Vaccine: Subjects vaccinated with cell-derived influenza vaccine.
Arm/Group | Egg-based Vaccine | Recombinant Vaccine | Cell-derived Vaccine
Number analyzed (Participants) | 4604 | 4614 | 4592
Participants
  SC2 Status | 131 | 157 | 141
  Influenza/SC2 Coinfection Status | 0 | 1 | 1

7. Other Pre Specified Outcome: Symptom Severity of SARS CoV2
Description: Symptom severity scores were reported by participants using FLU-PRO Plus (Influenza Patient Reported Outcomes), a standardized instrument developed to measure the intensity and frequency of viral respiratory tract symptoms. FluPRO Plus symptom scores range from 0 ("not at all") to 4 ("very much"), with higher scores indicating greater severity.
Time Frame: onset >13 days after Influenza vaccination up to 1 year
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Egg-based Vaccine: Subjects vaccinated with egg-based influenza vaccine.
- Recombinant Vaccine: Subjects vaccinated with recombinant influenza vaccine.
Arm/Group | Egg-based Vaccine | Recombinant Vaccine | Cell-derived Vaccine
Number analyzed (Participants) | 131 | 157 | 141
score on a scale | 1.00 [0.70 to 1.40] | 1.10 [0.70 to 1.50] | 1.10 [0.70 to 1.50]

ADVERSE EVENTS:
Time Frame: From study enrollment up to one year.
Arm/Group | Egg-based Vaccine | Recombinant Vaccine | Cell-derived Vaccine
All-Cause Mortality (participants affected / at risk) | 1/5145 | 1/5150 | 3/5137
Serious Adverse Events (participants affected / at risk) | 9/5145 | 5/5150 | 6/5137
Other Adverse Events (participants affected / at risk) | 0/5145 | 0/5150 | 0/5137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Egg-based Vaccine (N=5145) | Recombinant Vaccine (N=5150) | Cell-derived Vaccine (N=5137)
Hospitalization (General disorders) | 5 | 1 | 2
Hospitalization (Infections and infestations) | 1 | 3 | 3
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Hospitalization (Cardiac disorders) | 2 | 0 | 0
Hospitalization (Renal and urinary disorders) | 0 | 0 | 1
Hospitalization (Surgical and medical procedures) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-12-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT03734237/Prot_001.pdf
  • Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT03734237/SAP_002.pdf
  • Informed Consent Form (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT03734237/ICF_004.pdf